CLINICAL TRIAL: NCT00623792
Title: Preoperative Lifestyle Intervention in Bariatric Surgery
Brief Title: Study on Impact of Lifestyle Change and Weight Loss Before Bariatric Surgery
Acronym: PREP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duquesne University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Melissa Kalarchian, Associate Professor, Duquesne University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DK077102-01A1 (NIH); R01DK077102 (NIH)
Record Dates: First submitted 2008-02-14; First posted 2008-02-26 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Severe Obesity; Bariatric Surgery
Keywords: Morbid obesity; Diet therapy; Bariatric Surgery; Gastric bypass; Behavior therapy; Randomized controlled trial; Weight loss
MeSH Terms: conditions — Obesity, Morbid; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Usual preoperative care
- 2 (Experimental): Preoperative Lifestyle Intervention
  Interventions: Behavioral: Preoperative lifestyle Intervention

INTERVENTIONS:
Behavioral: Preoperative lifestyle Intervention — 6 month individual intervention consisting of weekly face-to-face and telephone sessions addressing diet, activity and preparation for surgery, followed by 3 "booster" telephone calls after surgery
  Arms: 2

SUMMARY:
The purpose of the trial is to determine whether a preoperative lifestyle intervention (targeting diet, exercise, and preparation for surgery) will favorably impact obesity-related parameters prior to bariatric surgery and improve short-term postoperative outcomes.

DETAILED DESCRIPTION:
This is a randomized, controlled trial to evaluate the impact of a preoperative lifestyle intervention that targets diet, exercise, and preparation for surgery as an adjunct to the surgical treatment of obesity. Patients will be randomized to a 6-month lifestyle intervention (n = 100) or to usual care (n = 100) prior to undergoing bariatric surgery. We aim to evaluate the effect of the intervention on select pre- and postoperative outcomes. We hypothesize that patients who participate in the preoperative intervention will exhibit greater improvements in weight and related outcomes and better preparation for surgery than those who receive usual care. After operation, we hypothesize that patients who participate in the intervention will exhibit better compliance and fewer behavior-related eating problems, as well as a lower rate of complications and fewer outpatient visits with surgery-related conditions than those who received usual preoperative care. Our secondary aim is to determine whether the intervention affects weight/BMI trajectory through 24 months after operation.

ELIGIBILITY:
Inclusion Criteria:

* Any candidate for weight loss surgery who is at least 18 years old [At the University of Pittsburgh Medical Center, bariatric surgery is recommended as a treatment for individuals with Class III obesity (BMI > 40), or Class II obesity (BMI 35- 40) and serious obesity-related health problems]

Exclusion Criteria:

* Mental retardation or psychosis
* Previously diagnosed genetic obesity syndrome
* Participation in a structured weight management program in the 6 months prior to study enrollment
* Uncontrolled psychiatric symptomatology sufficiently severe to require immediate treatment
* Pregnant or lactating in the previous 6 months
* Taking a medication known to affect body weight such as oral steroids in the previous 6 months
* Any previous surgery for weight loss
* Deemed high risk surgical candidate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2008-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
weight and related outcomes (BMI, cardiovascular risk, quality of life) | pre and post intervention
preparation for surgery (eating, activity and knowledge of surgery) | pre and post intervention
compliance and eating problems (vomiting, dumping, plugging etc.) | 6- and 12-months post surgery
surgical complications and outpatient visits | 6- and 12-months post surgery

SECONDARY OUTCOMES:
Weight/BMI trajectory | pre- and post-intervention; 6-, 12 and 24 months postop

CONTACTS AND LOCATIONS:
Overall Officials: Melissa A Kalarchian, PhD, Principal Investigator — Duquesne University
Locations (1):
- Duquesne University, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Kalarchian MA, Marcus MD, Courcoulas AP, Cheng Y, Levine MD. Self-report of gastrointestinal side effects after bariatric surgery. Surg Obes Relat Dis. 2014 Nov-Dec;10(6):1202-7. doi: 10.1016/j.soard.2014.08.007. Epub 2014 Aug 23. PMID 25443069